CLINICAL TRIAL: NCT07196592
Title: AD New Multi-Dimensional Therapy Device Development - Microcurrent Brain Stimulation Device and Virtual Reality Therapy Equipment
Brief Title: Development of a Novel Multidimensional Therapeutic Intervention Protocol for MCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuan Shen (Other)
Collaborators: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor-Investigator, Yuan Shen, MD., Ph.D., Tongji University
Organization: Tongji University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B20250001I
Record Dates: First submitted 2025-09-15; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: MCI-AD, Early Stage Alzheimer's Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Olfactory Stimulation Group (Experimental)
  Interventions: Behavioral: Olfactory stimulation
- TI Stimulation Group (Experimental)
  Interventions: Biological: Temporal Interference,TI
- Olfactory-TI Stimulation Group (Experimental)
  Interventions: Combination Product: Olfactory-TI Stimulation
- Sham Control Group (Sham Comparator)
  Interventions: Combination Product: Sham Control

INTERVENTIONS:
Behavioral: Olfactory stimulation — Olfactory stimulation were set as follows:
  Essential oil types: yuzu, lavender, lemon, and mint. Concentration: 158 μL of essential oil + 50 mL of water. The mixed solution was poured into the test tubes of the olfactory instrument, ensuring that the liquid levels of the four solutions were kept at the same height. Each scent was released for 30 seconds, followed by a 10-second air interval, with each cycle lasting 20 minutes.
  Arms: Olfactory Stimulation Group
Biological: Temporal Interference,TI — During stimulation, the parameters were set as follows:
  Δf=40Hz (2000Hz vs. 2040Hz) 2mA Stimulation duration: 20min We fixed the stimulation protocol and used a standard head to simulate stimulation of the entorhinal region.
  Arms: TI Stimulation Group
Combination Product: Olfactory-TI Stimulation — During stimulation, the parameters were set as follows:
  Δf=40Hz (2000Hz vs. 2040Hz) 2mA Stimulation duration: 20min We fixed the stimulation protocol and used a standard head to simulate stimulation of the entorhinal region.
  Olfactory stimulation were set as follows:
  Essential oil types: yuzu, lavender, lemon, and mint. Concentration: 158 μL of essential oil + 50 mL of water. The mixed solution was poured into the test tubes of the olfactory instrument, ensuring that the liquid levels of the four solutions were kept at the same height. Each scent was released for 30 seconds, followed by a 10-second air interval, with each cycle lasting 20 minutes.
  Arms: Olfactory-TI Stimulation Group
Combination Product: Sham Control — During stimulation, the parameters were set as follows:
  Δf=0Hz (2000Hz vs. 2000Hz) 2mA Stimulation duration: 20min.
  Olfactory stimulation were set as follows:
  Essential oil types: air. lasting 20 minutes.
  Arms: Sham Control Group

SUMMARY:
As populations age, Alzheimer's disease (AD) is increasing while disease-modifying drugs remain elusive, making early diagnosis and intervention essential. Building on advances in neuromodulation and virtual reality (VR), we target amnestic mild cognitive impairment (aMCI)-the prodromal stage of AD-as a key window for prevention. Preliminary evidence shows disrupted theta-delta phase-amplitude coupling in prefrontal and temporal cortices in aMCI, whereas olfactory enrichment can enhance hippocampal synaptic function, improve cognition, and potentially lower AD risk. We will conduct a large-scale clinical cohort study to test the neural mechanisms and clinical efficacy of multi-site, cross-frequency transcranial alternating current stimulation (tACS) combined with multisensory (visual-olfactory-auditory) VR. A comprehensive database spanning demographic, neuropsychological, biochemical, neuroimaging, and neuromodulation parameters will guide optimal protocols and provide objective evidence for non-pharmacological interventions, informing development of a microcurrent brain stimulator and a portable VR device.

DETAILED DESCRIPTION:
With the accelerating pace of population aging, the prevalence of Alzheimer's disease (AD) continues to rise, yet effective disease-modifying pharmacotherapies remain unavailable. Early diagnosis and intervention are critical to slowing cognitive decline and reducing disease burden. In recent years, rapid advances in neuromodulation and virtual reality (VR) have opened new avenues for mechanistic studies and functional brain rehabilitation in AD and other neurodegenerative disorders. Amnestic mild cognitive impairment (aMCI) is widely regarded as the prodromal stage of AD and represents a key window for prevention and treatment. Developing innovative non-pharmacological therapies for individuals at this early stage has therefore become an urgent clinical priority. Preliminary studies indicate that people with aMCI exhibit a significant loss of phase-amplitude coupling (PAC) between theta and delta rhythms in the prefrontal cortex and temporal lobe, whereas olfactory-enriched environmental stimulation can enhance hippocampal synaptic function, improve cognition, and lower AD risk. Accordingly, we propose a large-scale clinical cohort study to investigate the neural-circuit mechanisms and clinical efficacy of multi-site, cross-frequency transcranial alternating current stimulation (tACS) and multisensory VR integrating visual, olfactory, and auditory inputs for the treatment of aMCI. We will establish a comprehensive database encompassing demographic, neuropsychological, biochemical, neuroimaging, and neuromodulation parameters. Ultimately, this work will provide optimal theoretical parameters and objective evidence to guide the development of non-pharmacological interventions for AD-specifically, a microcurrent brain stimulator and a portable VR device.

ELIGIBILITY:
Inclusion Criteria:

Baseline screening inclusion criteria: a) Age ≤ 65 years and ≤ 85 years; b) Education duration ≥ 1 year; c) Normal cognitive function at enrollment: MMSE total score: non-illiterate (primary school or below) ≥ 20 points, primary school or above ≥ 24 points; d) Corrected vision and hearing are basically normal, and able to complete cognitive assessment.

Exclusion Criteria:

Baseline screening exclusion criteria: a) Neurological/psychiatric disorders affecting cognitive function: depression, schizophrenia, mental retardation, Parkinson's disease, etc.; b) Severe physical illnesses: cardiovascular disease, cerebrovascular disease, tumors, diabetes, kidney disease, and hypertension stage III or above; c) Autoimmune inflammatory diseases such as rheumatoid arthritis, lupus erythematosus, osteoarthritis, and multiple sclerosis.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Olfactory Sensitivity (TDI score) | Baseline; 30 minutes after Session 1; 30 minutes after Session 5; 30 minutes after Session 10; 1 week after Session 10.
  Change in olfactory function measured with the Sniffin' Sticks Threshold-Discrimination-Identification (TDI) composite score.
  Unit of Measure: TDI score, 1-48 (higher scores indicate better olfactory function).
Path Integration - Angle Deviation | Baseline; 5 minutes after Session 1; 5 minutes after Session 5; 5 minutes after Session 10.
  Absolute angular error during the path-integration task. Lower values indicate better performance.
  Unit of Measure: Degrees (°); lower is better.
Path Integration - Distance Deviation | Baseline; 5 minutes after Session 1; 5 minutes after Session 5; 5 minutes after Session 10.
  Difference between actual and ideal path length during the path-integration task. Lower values indicate better performance.
  Unit of Measure: Meters (m); lower is better.
Path Integration - Composite Accuracy (M_ROC_AUC) | Baseline; 5 minutes after Session 1; 5 minutes after Session 5; 5 minutes after Session 10.
  Area under the ROC curve computed from multivariate PI features to quantify task accuracy/reliability across sessions.
  Unit Measure: AUC, 0.00-1.00 (higher values indicate better accuracy/stability).
Change in Cognitive Performance (MoCA-B) | Baseline; 5 minutes after Session 10.
  Change in global cognition using the Montreal Cognitive Assessment-Basic (MoCA-B).
  Unit of Measure: MoCA-B score, 0-30 (higher scores indicate better cognition).

SECONDARY OUTCOMES:
Activities of Daily Living (ADL - Barthel Index) | Baseline; 30 minutes after Session 1; 30 minutes after Session 5; 30 minutes after Session 10; 1 week after Session 10.
  Change in functional ability using the Barthel Index. Unit of Measure: Barthel Index, 0-100 (higher scores indicate greater independence).
Adverse Events Related to Intervention | Baseline; 5 minutes after Session 1; 5 minutes after Session 5; 5 minutes after Session 10.
  Incidence of device- or procedure-related adverse events (e.g., skin irritation, headache, dizziness, nausea).
  Unit of Measure: Number of participants with ≥1 adverse event (count).

IPD SHARING:
Plan to Share IPD: No